CLINICAL TRIAL: NCT01003288
Title: Safety and Immunogenicity Studies of Pandemic Influenza (H1N1) 2009 Vaccine in Bergen
Brief Title: Studies of Pandemic Influenza (H1N1) 2009 Vaccine in Bergen
Acronym: H1N1VAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Cox, Professor, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H1N1VAC-2009, Version 1; 2009-016456-43 (EudraCT Number)
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: H1N1 pandemic vaccine immunogenicity safety; Health employees
MeSH Terms: interventions — pandemrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pandemic influenza H1N1 vaccine (Experimental): Influenza vaccine
  Interventions: Biological: Adjuvanted influenza H1N1split virion vaccine

INTERVENTIONS:
Biological: Adjuvanted influenza H1N1split virion vaccine — Vaccination Pandemrix suspension and emulsion for emulsion for injection. 1 dose (0.5 ml) contains Split influenza virus, inactivated, containing antigen 3.75 micrograms of A/California/7/2009 (H1N1)v-like strain (X-179A)
  * Pandemic influenza vaccine (H1N1)v (split virion, inactivated, adjuvanted)
  Other Names: Pandemrix

SUMMARY:
Haukeland University Hospital has approximately 8000 employees many of whom will be in the front line to receive the pandemic A/H1N1 vaccine. We propose to conduct a safety and immunogenicity study in these subjects

DETAILED DESCRIPTION:
The investigators will conduct a safety and immunogenicity study in health employees as detailed below:

* Examine adverse events of all employees after vaccination using adverse events form
* Examine the immunogenicity of the vaccine by collecting blood samples at days 0, 21 & 42 after vaccination (up to 500 people)
* Provide a detailed time course of the immune response to vaccination with a novel influenza H1N1 virus including the kinetics of the T-cell, B-cell and antibody responses in 50 volunteers
* Investigate the long lasting immunity induced by the vaccine
* Examine the ability of the vaccine to induce cross-reactive immunity to H1N1 strains.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent Subjects able to understand and comply with the study protocol and complete the Adverse Event Form Subjects able to attend the scheduled visits for the kinetic study

Exclusion Criteria:

* Persons with a history of anaphylaxis or serious reactions to any vaccine
* Person with known hypersensitivity to any of the vaccine components
* Persons who have had a temperature >38oC during the previous 72 hours
* Persons who have had an acute respiratory infection during the last 7 days
* Suspected non-compliance

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Espen Akselsen, MD, Study Chair — Haukeland University Hospital; Haakon Sjursen, MD PhD, Study Chair — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Result] Madhun AS, Akselsen PE, Sjursen H, Pedersen G, Svindland S, Nostbakken JK, Nilsen M, Mohn K, Jul-Larsen A, Smith I, Major D, Wood J, Cox RJ. An adjuvanted pandemic influenza H1N1 vaccine provides early and long term protection in health care workers. Vaccine. 2010 Dec 16;29(2):266-73. doi: 10.1016/j.vaccine.2010.10.038. Epub 2010 Oct 27. PMID 21034828
- [Result] Pedersen G, Halstensen A, Sjursen H, Naess A, Kristoffersen EK, Cox RJ. Pandemic influenza vaccination elicits influenza-specific CD4+ Th1-cell responses in hypogammaglobulinaemic patients: four case reports. Scand J Immunol. 2011 Aug;74(2):210-8. doi: 10.1111/j.1365-3083.2011.02561.x. PMID 21438900
- [Result] Jul-Larsen A, Madhun AS, Brokstad KA, Montomoli E, Yusibov V, Cox RJ. The human potential of a recombinant pandemic influenza vaccine produced in tobacco plants. Hum Vaccin Immunother. 2012 May;8(5):653-61. doi: 10.4161/hv.19503. Epub 2012 May 1. PMID 22634440
- [Result] Pathirana RD, Bredholt G, Akselsen PE, Pedersen GK, Cox RJ. A(H1N1)pdm09 vaccination of health care workers: improved immune responses in low responders following revaccination. J Infect Dis. 2012 Dec 1;206(11):1660-9. doi: 10.1093/infdis/jis589. Epub 2012 Sep 11. PMID 22969149
- [Result] Lartey S, Pathirana RD, Zhou F, Jul-Larsen A, Montomoli E, Wood J, Cox RJ. Single dose vaccination of the ASO3-adjuvanted A(H1N1)pdm09 monovalent vaccine in health care workers elicits homologous and cross-reactive cellular and humoral responses to H1N1 strains. Hum Vaccin Immunother. 2015;11(7):1654-62. doi: 10.1080/21645515.2015.1048939. PMID 26009966
- [Result] Eidem S, Tete SM, Jul-Larsen A, Hoschler K, Montomoli E, Brokstad KA, Cox RJ. Persistence and avidity maturation of antibodies to A(H1N1)pdm09 in healthcare workers following repeated annual vaccinations. Vaccine. 2015 Aug 7;33(33):4146-54. doi: 10.1016/j.vaccine.2015.05.081. Epub 2015 Jun 7. PMID 26057137
- [Result] Trieu MC, Zhou F, Lartey SL, Sridhar S, Mjaaland S, Cox RJ. Augmented CD4+ T-cell and humoral responses after repeated annual influenza vaccination with the same vaccine component A/H1N1pdm09 over 5 years. NPJ Vaccines. 2018 Aug 14;3:37. doi: 10.1038/s41541-018-0069-1. eCollection 2018. PMID 30131880
- [Result] Trieu MC, Zhou F, Lartey S, Jul-Larsen A, Mjaaland S, Sridhar S, Cox RJ. Long-term Maintenance of the Influenza-Specific Cross-Reactive Memory CD4+ T-Cell Responses Following Repeated Annual Influenza Vaccination. J Infect Dis. 2017 Mar 1;215(5):740-749. doi: 10.1093/infdis/jiw619. PMID 28007925
- [Result] Trieu MC, Jul-Larsen A, Saevik M, Madsen A, Nostbakken JK, Zhou F, Skrede S, Cox RJ. Antibody Responses to Influenza A/H1N1pdm09 Virus After Pandemic and Seasonal Influenza Vaccination in Healthcare Workers: A 5-Year Follow-up Study. Clin Infect Dis. 2019 Jan 18;68(3):382-392. doi: 10.1093/cid/ciy487. PMID 29893797
- [Derived] Amdam H, Madsen A, Zhou F, Bansal A, Trieu MC, Cox RJ. Functional and Binding H1N1pdm09-Specific Antibody Responses in Occasionally and Repeatedly Vaccinated Healthcare Workers: A Five-Year Study (2009-2014). Front Immunol. 2021 Dec 6;12:748281. doi: 10.3389/fimmu.2021.748281. eCollection 2021. PMID 34938285
- [Derived] Manenti A, Tete SM, Mohn KG, Jul-Larsen A, Gianchecchi E, Montomoli E, Brokstad KA, Cox RJ. Comparative analysis of influenza A(H3N2) virus hemagglutinin specific IgG subclass and IgA responses in children and adults after influenza vaccination. Vaccine. 2017 Jan 3;35(1):191-198. doi: 10.1016/j.vaccine.2016.10.024. Epub 2016 Oct 24. PMID 27789145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HCW working at Haukeland University Hospital during the influenza pandemic in 2009
Groups:
- Pandemic Influenza Vaccine (H1N1)v: Pandemrix: Vaccination Pandemrix suspension and emulsion for emulsion for injection. 1 dose (0.5 ml) contains Split influenza virus, inactivated, containing antigen 3.75 micrograms of A/California/7/2009 (H1N1)v-like strain (X-179A)
  * Pandemic influenza vaccine (H1N1)v (split virion, inactivated, adjuvanted)
Period: Overall Study
Arm/Group | Pandemic Influenza Vaccine (H1N1)v
Started | 255
Completed | 255
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Health Care Workers: Received one or two doses of pandemic vaccine during 2009 pandemic and susbequent seasonal vaccination was optional
- Hypogammaglobulinaemic Patients: Received two doses of pandemic vaccine
- Total: Total of all reporting groups
Arm/Group | Health Care Workers | Hypogammaglobulinaemic Patients | Total
Number analyzed (Participants) | 251 | 4 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 251 | 4 | 255
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 3 | 198
  Male | 56 | 1 | 57
Region of Enrollment [Number; unit: participants]
  Norway | 251 | 4 | 255

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Adverse Events
Description: Solicited adverse events were collected on side reactions form which were filled in for 21 days after pandemic or seasonal vaccination.
Time Frame: 21 days after vaccination
Population: solicited adverse event forms were collected from the volunteers
Measure: Number; unit: participants
Groups:
- Pandemic Vaccine: Pandemic Vaccine in HCW
Arm/Group | Pandemic Vaccine
Number analyzed (Participants) | 255
participants | 207

2. Secondary Outcome: Number of Participants With Immunogenicity as Determined Using Haemagglutination Inhibition Assay
Description: Antibody responses were measured using the HI assay to evaluate the rapidity and long term duration of the response
Time Frame: 7, 14, 21 days post vaccination and long term follow up for 5 years
Population: Only HCW 251 were assessed for HI antibodies at 21 days post vaccination
Measure: Number; unit: participants
Arm/Group | HCW Pandemic Vaccine
Number analyzed (Participants) | 251
participants | 251

ADVERSE EVENTS:
Time Frame: 5 year follow up
Groups:
- Pandemic Vaccine: HCW vaccinated with pandemic vaccine
Arm/Group | Pandemic Vaccine
Serious Adverse Events (participants affected / at risk) | 0/255
Other Adverse Events (participants affected / at risk) | 196/255
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pandemic Vaccine (N=255)
pain at injection site (Infections and infestations) | 196 (196)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes